CLINICAL TRIAL: NCT00190177
Title: ECLAXIR:Search for an Association Between CX3CR1 V249I Polymorphism, Preeclampsia and Endothelial Injury
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: P020925
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2013-10-18 (Estimated); Status verified 2005-09

CONDITIONS: Preeclampsia
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The study hypothesis is the involvement of the couple CX3CR1/CX3CL1 in occurrence of endothelial injury in preeclampsia. According to this hypothesis, Carriers of the I249 allele who express less CX3CR1 shoud be protected against this risk. The main objective of the study is the search of an association between CX3CR1 V249I polymorphism and preeclampsia. The secondary aims are the search of an association with the most severe forms of preeclampsia and endothelial injury.

DETAILED DESCRIPTION:
It is a case-control multicenter study 185 caucasian pregnant women with preeclampsia and 185 paired controls without preeclampsia will be included.

The frequency of the V249I polymorphism in african black population will be determined by studying 200 subjects (100 cases and 100 controls).

The V249I polymorphism will be identified by PCR followed by enzyme digestion. Endothelial injury will be identified using three assays : von Willebrand factor, soluble VCAM-1 and thrombomodulin plasma levels.

CX3CR1 involvement in preeclampsia would have potential diagnostic and therapeutic consequences.

ELIGIBILITY:
Inclusion Criteria:

* cases: pregnant woman, evolutive pregnancy, preeclampsia, caucasian, consenting to the study

Exclusion Criteria:

* Cases:

multiple pregnancy, proteinuria > 300 mg/24h before 21th gestation week.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 370 (Estimated)
Dates: Start 2003-03; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laurent Mandelbrot, MD-PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Louis Mourier AP-HP, Colombes, France